CLINICAL TRIAL: NCT06116448
Title: The Effectiveness of Simulation-Based Education on Nursing Students' Breastfeeding Knowledge, Skills, Confidence, and Satisfaction.
Brief Title: Nursing Students& Breastfeeding Education& Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, sümeyye bakır, doctoral student/research assistant, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: E.496527
Record Dates: First submitted 2023-10-23; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Breastfeeding
Keywords: breastfeeding; nursing students; Nursing Research, Educational
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: prospective, parallel, randomized, controlled quasi-experiment
Who Masked: Participant
Masking Description: The students who participated in the research were unaware of which group they were assigned to and attended the practices accordingly. During the clinical follow-up phase, a clinical breastfeeding nurse evaluated the practices using a checklist but did not know which group the students belonged to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- high-fidelity simulation (Experimental): These students participated in a breastfeeding management scenario with a high-fidelity simulation mannikin named Noella S554.100 (n=11).
  Interventions: Other: high-fidelity simulation
- hybrid simulation (Experimental): These students participated in the same breastfeeding management scenario with a standardized patient (n=11).
  Interventions: Other: hybrid simulation
- telesimulation (Experimental): These students participated in the same breastfeeding management scenario with a standardized patient via Microsoft Teams video conferencing. (n=11)
  Interventions: Other: telesimulation
- control (No Intervention): The students in this group were the control group, and no intervention was made.

INTERVENTIONS:
Other: high-fidelity simulation — The high-fidelity simulation involved a student and a computer-based mannikin. Prior to the start of the scenario, a pre-briefing session was provided. The scenario was executed with the help of the researcher from the control room. The student's performance during the simulation was recorded with video. Each simulation lasted around 30 minutes. Following the simulation, a debriefing session was held with the student, and feedback was provided. Scales were used to assess the implementation of the practices.
  Arms: high-fidelity simulation
Other: hybrid simulation — The hybrid simulation involved a student and a standardized patient. The patient wore a wearable breast model and held a model baby. Prior to the start of the scenario, a pre-briefing session was provided. The student's performance during the simulation was recorded with video. Each simulation lasted around 30 minutes. Following the simulation, a debriefing session was held with the student, and feedback was provided. Scales were used to assess the implementation of the practices.
  Arms: hybrid simulation
Other: telesimulation — The telesimulation involved a student and a standardized patient. The patient wore a wearable breast model and held a model baby. Students and patients communicated via video conferencing. Prior to the start of the scenario, a pre-briefing session was provided. The student's performance during the simulation was recorded with video. Each simulation lasted around 30 minutes. Following the simulation, a debriefing session was held with the student, and feedback was provided. Scales were used to assess the implementation of the practices.
  Arms: telesimulation

SUMMARY:
The study aimed to determine the effect of different simulation methods on nursing students' self-confidence, satisfaction, and clinical breastfeeding management knowledge and skills in managing and supporting breastfeeding in the early postpartum period.

DETAILED DESCRIPTION:
This study aimed to investigate the effectiveness of simulation-based training methods in improving the breastfeeding management knowledge and skills of third-year nursing students. The study utilized a quasi-experimental design with pre-test and post-test control groups. The results of the intervention groups that received high-fidelity, hybrid, and telesimulation training were compared with a control group that received traditional training. A clinical follow-up phase was conducted after the interventions to evaluate their impact. The study used various data collection tools to measure different factors, including knowledge and skills, confidence in learning, satisfaction, training satisfaction, and self-assessment of simulations.

ELIGIBILITY:
Inclusion Criteria:

The voluntarily agree to participate in the study Not having experience with simulation Being a 3rd year nursing undergraduate student not working as a nurse

Exclusion Criteria:

During the study, participants must complete all forms, attend all theoretical training, and remain in the study until completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
breastfeeding management knowledge | change from before implemention and 5th week of after practice
  The researchers developed a measurement tool to assess information. The tool uses a scoring system where correct statements receive one point and incorrect statements receive zero points. The total score ranges from 0 to 47 points.
breastfeeding management skills | through simulation practices completion, an average of 5 weeks and through clinical practices completion, an average of 5 weeks
  The researchers developed a checklist to assess skills. The tool uses a scoring system where correct practice receives one point and incorrect statements receive zero points. The checklist consists of seven sections. The number of items in each section ranges from 4 to 14.
Evaluation of Breastfeeding Education | change from before implemention and 5th week of after practice
  The researchers developed a measurement tool to assess breastfeeding education. The form items are evaluated as feeling adequate or inadequate (1 or 0 points). The total score ranges from 0 to 27 points.

SECONDARY OUTCOMES:
students' self-confidence and satisfaction | through simulation practices completion, an average of 5 weeks
  It is a scale published by the National League for Nurses (NLN) to measure students' attitudes and beliefs about simulation.The highest score that can be obtained from the scale is 65 and the lowest score is 13.
self-evaluation | through simulation practices completion, an average of 5 weeks
  The self-report scale assesses the impact of simulation lab practices on nursing students' professional knowledge, skills, and attitudes.The lowest score that can be obtained from the scale is 0 and the highest score is 92.
education methods satisfaction | through simulation practices completion, an average of 5 weeks and through clinical practices completion, an average of 5 weeks
  It evaluates the degree of contentment of the student with the teaching methodology implemented.In evaluating the satisfaction with training methods, students are scored from 20 to 80.

CONTACTS AND LOCATIONS:
Overall Officials: sümeyye bakır, master, Principal Investigator — Ege University
Locations (1):
- Sümeyye Bakır, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The researchers intend to publish the study as an article
Supporting Information: Study Protocol
Time Frame: from January 2025
Access Criteria: the article is planned to be published as open access

REFERENCES:
- [Background] Sittner BJ, Aebersold ML, Paige JB, Graham LL, Schram AP, Decker SI, Lioce L. INACSL Standards of Best Practice for Simulation: Past, Present, and Future. Nurs Educ Perspect. 2015 Sep-Oct;36(5):294-8. doi: 10.5480/15-1670. PMID 26521497
- [Background] Toruner EK, Altay N, Arpaci T, Sari Ozturk C, Ceylan C, Yildiz S, Cakir G. The development of a self-evaluation scale for simulation laboratory practices. Nurse Educ Today. 2021 Sep;104:104990. doi: 10.1016/j.nedt.2021.104990. Epub 2021 Jun 2. PMID 34146847
- [Background] Moloney M, Murphy L, Kingston L, Markey K, Hennessy T, Meskell P, Atkinson S, Doody O. Final year undergraduate nursing and midwifery students' perspectives on simulation-based education: a cross-sectional study. BMC Nurs. 2022 Nov 6;21(1):299. doi: 10.1186/s12912-022-01084-w. PMID 36335322